CLINICAL TRIAL: NCT04828525
Title: Corticosteroids as an Additional Treatment for Mastoiditis In Children
Acronym: COSMIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ori snapiri (Other)
Responsible Party: Sponsor-Investigator, ori snapiri, Pediatrician, Principal Investigator, Clinical doctor, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0702-20-RMC
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Mastoiditis; Acute
Keywords: mastoiditis; children; corticosteroids
MeSH Terms: conditions — Mastoiditis | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Intervention Model Description: The research is a multi-centered, prospective, placebo-control, randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: participants will be randomized divided into two groups. each group will be given dexamethasone or 0.9% normal saline. only the pharmacist will not be masked to the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): participants will be given corticosteroids in addition to conventional treatment
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): participants will be given normal saline in addition to conventional treatment
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexamethasone — adjuvant dexamethasone treatment
  Arms: Experimental
Drug: normal saline — placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the influence of adjuvant corticosteroid treatment in acute mastoiditis in children. we expect a better outcome in children treated with both corticosteroids and antibiotics including lower rates in complications and earlier decline in fever and inflammatory markers.

DETAILED DESCRIPTION:
The research is a multi-centered, prospective, placebo-control, randomized controlled trial. The study group will be comprised of children diagnosed with acute mastoiditis and hospitalized in a pediatric medical center.

The participating patients will be randomized divided into two groups. Research group will be given dexamethasone treatment (course of 16 doses, 0.15 mg/kg/dose every 6 hours) in addition to antibiotic treatment. Control group will be given 16 doses of 0.9% normal saline in addition to antibiotic treatment. Management and treatment will be conducted according to clinical condition and laboratory findings as for routine institution protocols. It should be noted that the regular institutional management of children enrolled for the study will not be changed due to our research.

ELIGIBILITY:
Inclusion Criteria:

* acute mastoiditis

Exclusion Criteria:

* immunodeficiency (congenital or acquired)
* significant chronic disease
* hypertension
* recurrent mastoiditis

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Time from the beginning of the treatment until clinical and laboratory findings are within normal limits | during hospitalization, anticipated 1-2 weeks
  fever, crp levels

SECONDARY OUTCOMES:
Complication rates | during hospitalization, anticipated 1-2 weeks
  sinus vein thrombosis, intracranial collection or abscess, need for surgery

OTHER OUTCOMES:
Duration of hospitalization | anticipated 1-2 weeks
  time from admission until discharge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin HW, Shargorodsky J, Gopen Q. Clinical strategies for the management of acute mastoiditis in the pediatric population. Clin Pediatr (Phila). 2010 Feb;49(2):110-5. doi: 10.1177/0009922809344349. Epub 2009 Sep 4. PMID 19734439
- [Background] Groth A, Enoksson F, Hultcrantz M, Stalfors J, Stenfeldt K, Hermansson A. Acute mastoiditis in children aged 0-16 years--a national study of 678 cases in Sweden comparing different age groups. Int J Pediatr Otorhinolaryngol. 2012 Oct;76(10):1494-500. doi: 10.1016/j.ijporl.2012.07.002. Epub 2012 Jul 23. PMID 22832239
- [Background] Delgado-Noguera MF, Forero Delgadillo JM, Franco AA, Vazquez JC, Calvache JA. Corticosteroids for septic arthritis in children. Cochrane Database Syst Rev. 2018 Nov 21;11(11):CD012125. doi: 10.1002/14651858.CD012125.pub2. PMID 30480764
- [Background] Aljebab F, Choonara I, Conroy S. Systematic review of the toxicity of short-course oral corticosteroids in children. Arch Dis Child. 2016 Apr;101(4):365-70. doi: 10.1136/archdischild-2015-309522. Epub 2016 Jan 14. PMID 26768830
- [Background] Brouwer MC, McIntyre P, Prasad K, van de Beek D. Corticosteroids for acute bacterial meningitis. Cochrane Database Syst Rev. 2015 Sep 12;2015(9):CD004405. doi: 10.1002/14651858.CD004405.pub5. PMID 26362566